CLINICAL TRIAL: NCT06380920
Title: Function Definition and Clinical Validation of Digital Health App: Using Weight Management as An Example
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chih-Hsing Wu, Professor, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Digital Health App
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-05

CONDITIONS: Weight Loss; Body Fat Rate Loss; Body Composition Change
Keywords: obesity; assistive intelligence; APP; weight control; cognitive behavior therapy
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case (Experimental): intervened with App/CBT/MB-EAT groups by a randomized control trial design for 9 months and periodically surveyed as well as 0, 3, and 6 months after intervened
  Interventions: Device: "AI Mindful Eating" App; Behavioral: Outpatient regular follow-up
- Control (Placebo Comparator): intervened without App/CBT/MB-EAT groups by a randomized control trial design for 9 months and periodically surveyed as well as 0, 3, and 6 months after intervened
  Interventions: Behavioral: Outpatient regular follow-up

INTERVENTIONS:
Device: "AI Mindful Eating" App — The investigators propose on design of an "AI Mindful Eating" App, to enhance individual's healthy lifestyle with subsequent weight-loss. Based on "gut-brain axis," this is anticipated to be achieved by using CBT, in place of medication, to alleviate food addiction and proper nutrition intake during proper metabolic conditions and time, which are coordinated via AI.
  Arms: Case
Behavioral: Outpatient regular follow-up — Outpatient regular follow-up

SUMMARY:
This project anticipates addressing the obesity epidemics problem which has caused unhealthy lifestyle in billions of obesities and overweight people worldwide. The investigators propose on digital health solution in providing healthcare-on-demand, for personalized health, healthy lifestyle and weight management. This study proposes on using Cognitive Behavior Therapy (CBT) in decreasing individual's food craving, which is administered through AI (Assistive Intelligence) tracking. As with any new medicine, uncertain long-term effects and high costs of these new drugs are also critical factors considered by physicians and policy makers worldwide. Researchers have also reported on 85% of people re-gaining premedication weight after 5 years. There is no easily available self-controlled monitoring strategy/intervention for the unhealthy lifestyle is believed to be one of the main problems. Therefore, the investigators propose on the research and development of self-managing digital health APP (application) for 12 months over two phases, with three months to design APP and nine months to confirm the clinical validation. During the first phase, the investigators propose on design of an "AI Mindful Eating" App, to enhance individual's healthy lifestyle with subsequent weight-loss. Based on "gut-brain-axis", this is anticipated to be achieved by using CBT and AI is used to recognize nutrition and mood within mobile images. This facilitates fulfilling lifestyle and long-term weight-loss. Finally, the study proposes to complete function definition and clinical validation for our AI Humanity APP. By scheduled check-up program by monitoring and analyzing body weight, body fat, anthropometric and metabolic change data between case and control groups. The investigators intend to disclose the effect of the AI assistant APP in weight management and metabolic disease prevention.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects (BMI>= >= 27 kg/m2) with age 18 year-old and less than 65 y/o over will be considered (M/F= 1:1)

Exclusion Criteria:

* Any history of cancer
* Unstable mental status
* Uncooperative subject
* Complex clinical comorbidities, such as heart failure, end-stage renal disease, etc.
* Severe physical disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
weight change | 0, 3 and 6 months after intervened
  Body composition measured by BIA or DXA

SECONDARY OUTCOMES:
Parameters of Metabolic syndrome | 0, 3 and 6 months after intervened
  Waist circumference was measured at mid-way of abdomen during end-expiratory phase

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hsing Wu, MD, Study Director — Department of Family Medicine, National Cheng Kung Univ Hosp
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No